CLINICAL TRIAL: NCT02948153
Title: Asthma With Bronchial Hypersecretion: Expression of Mucins and Toll-like Receptors in Sputum and Blood
Brief Title: Mucins and Toll-like Receptors in Asthma
Acronym: MUCITOLL
Status: Completed | Type: Observational
Sponsor: Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau (Other)
Collaborators: Spanish Respiratory Society (Other)
Responsible Party: Sponsor
Other Study IDs: IIBSP-ROF-2011-106
Record Dates: First submitted 2016-10-18; First posted 2016-10-28 (Estimated); Last update posted 2016-10-28 (Estimated); Status verified 2015-09

CONDITIONS: Asthma; Inflammation
MeSH Terms: conditions — Asthma; Inflammation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- asthma with bronchial hypersecretion: In a clinical study, participants are often divided into groups. Group one: they were defined as those who expectorated daily for at least three months for a minimum period of two consecutive years, without attribution to any other cause or disease.
  Interventions: Other: clinical study
- asthma without hypersecretion: In a clinical study, participants are often divided into groups. Group two: We defined asthma as a history of variable respiratory symptoms and evidence of variable expiratory airflow limitation.
  Interventions: Other: clinical study

INTERVENTIONS:
Other: clinical study — It is a comprehensive study in a large sample using multiple techniques to assess various aspects of the disease. All patients underwent the following : Induced Sputum, spirometry, fractional exhaled nitric oxide (FeNO), prick test, total IgE and blood albumin. Analysis of mucins and TLRs

SUMMARY:
This study raises two main hypotheses: 1) Asthmatics patients who present with bronchial hypersecretion differ phenotypically from asthmatic patients without hypersecretion and 2) mucins in asthmatic patients with hypersecretion of bronchial mucus and the expression of TLRs differ from non-mucus hypersecretory asthmatics patients.

DETAILED DESCRIPTION:
Asthma with bronchial hypersecretion is a type of asthma poorly studied. Its pathogenesis is not well understood but probably is related to the innate impaired immunity, particularly with "toll-like receptors" (TLR) and secretory mucin (MUC).

Objectives 1) Define the clinical and inflammatory phenotype of asthma with bronchial hypersecretion of mucus. 2) Compare the type of mucin present in induced sputum (IS) of patients with and without bronchial hypersecretion. 3) Determine the expression of TLRs in the IS and in the peripheral blood of asthmatics with and without bronchial hypersecretion.

Method: Cross-sectional study which included 43 asthmatic patients, 19 with and 24 without bronchial hypersecretion. All patients underwent the following: IS, spirometry, fractional exhaled nitric oxide (FeNO), prick test, total IgE and blood albumin. Analysis of mucins (MUC2, MUC5AC, MUC5B and MUC1) was determined by ELISA and expression of TLR2 and TLR4 by flow cytometry. The level of asthma control was determined by the asthma control test questionnaire (ACT) and quality of life was assessed by the MiniAQLQ questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* Non-smokers, asthma diagnosed as per the Global INitiative for Asthma (GINA) criteria on maintenance treatment for asthma, aged 18 to 80 years.

Exclusion Criteria:

* Patients were excluded from the study if they had a respiratory tract infection and/or required the use of oral corticosteroids within 30 days prior to inclusion; if they had a concomitant disease (sarcoidosis, lung cancer, pulmonary tuberculosis, bronchiectasis, nephropathy, rheumatic or liver disease); significant comorbidity that could affect the study results in the physician's judgment; or a cognitive impairment that could limit their comprehension of the subject under study or their ability to participate

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Male and female subjects aged > 18 years, non-smokers, who fulfilled the diagnostic criteria of asthma were consecutively enrolled from the Asthma Unit outpatient clinic of our institution. We defined asthma as a history of variable respiratory symptoms and evidence of variable expiratory airflow limitation. All patients had a positive bronchodilator test or daily peak expiratory flow variability greater than 20%, or a positive methacholine challenge test documented in case history. Asthma severity was defined according to the Global Initiative for Asthma Management (GINA)
Sampling Method: Probability Sample
Enrollment: 43 (Actual)
Dates: Start 2014-01; Primary Completion 2015-09 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Number of asthmatic patients with bronchial hypersecretion | 18 months

SECONDARY OUTCOMES:
Number of asthmatic patients with altered expression of TLRs | 18 months
Number of asthmatic patients with altered expression of Mucins | 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Astrid Crespo, MD,PHD, Principal Investigator — Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau
Locations (1):
- Hospital de la Santa Creu i Sant Pau. Carrer Mas Casanovas 90., Barcelona, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No